CLINICAL TRIAL: NCT03367507
Title: The Effect of Individually Tailored Sub-maximal Exercise Prescription in Adolescent Physiological Post-concussion Disorder: a Multi-institutional Randomized Controlled Trial
Brief Title: Sub-maximal Exercise Prescription in Adolescents With Physiological Post-concussion Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sport Injury Prevention Research Centre (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB17-0570
Record Dates: First submitted 2017-11-16; First posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Physiological Post-Concussion Disorder; Post-Concussion Syndrome; Traumatic Brain Injury; Rehabilitation; Aerobic Exercise; Concussion, Brain
MeSH Terms: conditions — Post-Concussion Syndrome; Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Intervention Model Description: Research statement:This study is a multi-centre RCT. The purpose of the RCT is to evaluate the efficacy of a moderate intensity (80% symptom threshold HR, Borg RPE 12-16) sub-symptom aerobic exercise prescription compared to a lower level aerobic exercise group (60% HR, Borg RPE 7-11) on time to medical clearance to receive medical clearance to return to play in adolescents (aged 13-19) with suggested physiological Post-Concussion Disorder (P-PCD).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not be blinded to group assignment, as it would be impossible to make them unaware of how intense their exercise prescription should be but they will be blinded to the other treatment assignment and masked to the study hypothesis. The treating sport medicine physician will be blinded to group assignment. There will be an exercise physiologist who will be responsible for conducting the treadmill tests and, prescribing aerobic exercise programs. The study exercise physiologist will not be blinded and will not relay any information pertaining to group assignment to other members involved in the study other than the participants themselves and their parents. Those assessing adverse events will not be masked and if needed to facilitate clinical care the managing physician will be made aware of the treatment group. Compliance will be tracked through the use of Actigraph accelerometers, heart rate monitors and daily activity logs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 80% Sub-symptom threshold aerobic exercise (Experimental): The moderate intensity intervention group will exercise at 80% of the maximum symptom free heart rate identified by their most recent graded treadmill test. The target heart rate zone will be within of the heart rate at which they experienced an increase in symptoms. The participants will be instructed to follow a program of moderate intensity activity in the form of their choice, we will recommend the following: stationary cycling, brisk walking, light jogging or the use of any available cardiovascular exercise equipment where they can control and monitor their heart rate wearing both the Actigraph and Polar HR monitor provided.
  Interventions: Behavioral: Sub-symptom aerobic exercise
- 60% Sub-symptom aerobic exercise (Active Comparator): The light (conservative) intensity intervention group will exercise at 60% of the maximum symptom free heart rate identified by their most recent graded treadmill test. The target heart rate zone will be within of the heart rate at which they experienced an increase in symptoms. The low intensity group will perform their exercise program at their own discrepancy however we will advise either of the following activities: light walking, stationary cycling or the use of any available cardiovascular exercise equipment where they can control and monitor their heart rate while simultaneously wearing both the Actigraph and polar HR monitor.
  Interventions: Behavioral: Sub-symptom aerobic exercise

INTERVENTIONS:
Behavioral: Sub-symptom aerobic exercise — Both groups will be instructed to perform their respective aerobic exercise program the following day after completing their first treadmill test. Participants will be instructed to exercise at their prescribed intensity for a maximum of 30 minutes a day, 4-5 days a week. They will be asked to postpone the exercise until the next day if they experience significant increases in symptoms from usual resting levels. Exercise type will be the participant's choice, however we will ask the participant refrain from contact/high risk activities including any modalities that might induce rapid and aggressive head movements.

SUMMARY:
Although the vast majority of individuals sustaining a sport-related concussion (SRC) will receive medical clearance to return to sport within 7-10 days, approximately 30% of children and adolescents reporting to the emergency department will experience symptoms that last longer than a month. Research has demonstrated that exercise below the threshold that results in increases in symptoms, beyond those experienced at rest, (sub-symptom threshold aerobic exercise) may be beneficial in recovery. However, the optimal amount and intensity of aerobic exercise for an individual to experience the most beneficial outcomes is currently unknown. Unfortunately there are limited Randomized Controlled Trials (RCT's) evaluating the benefits of aerobic exercise in a youth population. The current evidence includes studies with relatively small sample sizes, unreliable measurements of physical activity (self-report), and inherent biases through inadequate blinding. There is a need to develop and validate evidence-informed interventions as a means of treatment for limiting time loss from sport, and school in adolescents who experience persistent symptoms of sports related concussion beyond 10 days.

DETAILED DESCRIPTION:
Research statement:This study is a multi-centre RCT. The purpose of the RCT is to evaluate the efficacy of a moderate intensity (80% symptom threshold heart rate (HR), Borg Rating of Perceived exertion (RPE) 12-16) sub-symptom aerobic exercise prescription compared to a conservative low level aerobic exercise group (60% HR, Borg RPE 7-11) on time to medical clearance to return to play in adolescents (aged 13-19) with suggested physiological Post-Concussion Disorder (P-PCD).

Secondary objectives are to 1) Measure the adherence patterns of youth who are prescribed a specific aerobic home exercise programs. 2) Monitor longitudinal symptom reduction on the Sport Concussion Assessment Tool 5 (SCAT5) (week 0 and medical clearance) 3) Track longitudinal changes in patient-reported outcomes (symptoms) through the use of the Pediatric Quality of Life (PedsQL) questionnaire. 4) Evaluate the association between cognitive activity and time to receive medical clearance to return to sport.

Methods: A multisite RCT will be conducted at the Pan Am Concussion Program, Winnipeg, Manitoba and the Sport Injury Prevention Research Centre/Acute Sport Concussion Clinic, Sport Medicine Centre, Faculty of Kinesiology, University of Calgary, Calgary, Alberta. Adolescents (n=136, 68 from each study site, ages 13-19 years) who are diagnosed with a sport-related concussion and have ongoing symptoms for more than 10 days but less than 30 days will be recruited for study participation. Participants will be randomized via permuted block to either a moderate intensity (80%) or a low intensity (60%) aerobic exercise intervention. Both groups will be instructed to perform their respective home aerobic exercise program the beginning the day after completing their first treadmill test. Participants will be instructed to exercise at their prescribed intensity for a maximum of 30 minutes a day, 4-5 days a week. In the unlikely event in which participants feel unable to continue their home exercise program they will be asked to postpone the exercise until the next day. Participants will undergo diagnostic treadmill tests every two weeks, which will be used to determine increases in exercise tolerance and serve as a parameter of physiological recovery. The treadmill tests will also be used to set a new threshold heart rate for a person to continue to exercise at for the following two weeks or until receiving medical clearance to initiate the return to play protocol. The treadmill test is made to represent the most similar form of exercise to mimic an adolescent's respective sport.

Participants will also be asked to fill out the SCAT5 symptom scores before and after treadmill testing along with the PedsQl questionnaire. Self-reported physical and cognitive activity will be tracked with daily exercise logs, these will be used in conjunction with Actigraph accelerometers and heart rate monitors which will serve as objective tools to track the quantification of physical activity.

Data safety and monitoring: The study team at the University of Manitoba have performed over 200 treadmill tests in a pediatric concussed population with no challenges regarding safety or tolerability. The study staff will be qualified to perform exercise stress tests in a safe manner based on standards of practice imposed by the University of Calgary and Canadian Society for Exercise Physiology. All study practices will be conducted under the supervision of a physician and exercise physiologist who are trained at a minimum level of cardio pulmonary resuscitation (CPR) level C and trained to use an automated external defibrillator (AED). All study personnel will know the location and how to use the on-site AED's. Monthly teleconferences will be held between the research team at the University of Manitoba and University of Calgary regarding, safety, logistics and proper manners in which to conduct exercise tests. Between both sites we will establish a data safety and monitoring committee to ensure the safety of all patients. This independent group of experts will monitor patient safety and treatment efficacy during the ongoing RCT and report their findings to the primary investigators. The committee's role will be to periodically review and evaluate the data collected thus far for any concerns related to patient safety or study conduct. If needed, they will also provide recommendations about the continuation, modification, or termination of the RCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-19 years
2. Physician diagnosed sports-related concussion, defined according to the 5th International Consensus Statement on Concussion in Sport (McCrory et al., 2017) as an injury caused by transmission of biomechanical forces to the brain leading to clinical symptoms affecting multiple domains of physical, cognitive, sleep, and neurobehavioral functioning (McCrory et al., 2017);
3. persistent symptoms at 10-30 days post-concussion;
4. a post-concussion symptom scale score greater than 5 for males and 8 for females (these are above the typically reported values for non-concussed athletes);
5. self reported difficulties with exertion and/or a graded aerobic treadmill test demonstrating isolated Physiological Post Concussion Disorder;
6. participant and parent/guardian informed consent;
7. Participant must be able to reach a heart rate greater than 100 but less than 210 bpm, during and throughout the onset of exercise (to ensure their sub-symptom threshold is still above resting norms);
8. Voluntary consent to wear an Actigraph (wGT3X-BT) accelerometer monitor for a minimum of 2 weeks and the provided Polar HR monitor during daily exercise.

Exclusion Criteria:

1. clinical evidence of vestibulo-ocular dysfunction (Ellis, et al., 2015; 2017);
2. clinical evidence of cervical spine soft tissue injury (Schneider et al., 2014);
3. past medical history of International Classification of Diseases-3 beta version migraine headaches;
4. undergoing active medical treatment for a psychiatric disorder (e.g. on medication for depression);
5. contraindication to exercise testing (traumatic abnormality on neuroimaging studies, co-existing cardiac, respiratory or orthopedic contraindication to exercise testing, pregnancy);
6. exercise intolerance reached before 100 bpm, or after 210 bpm (age predicted maximum heart rate) on graded exercise test;
7. subjects refusal to wear Actigraph and Polar HR monitor;
8. subjects resting HR above 99bpm or blood pressure greater than 144/94.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 136 (Estimated)
Dates: Start 2017-12-10 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Days to receive medical clearance to return to sport | up to 8 weeks
  The time it takes in days for the physician to provide clearance to the participant to return to sport (calculated from date of initiation of intervention)

SECONDARY OUTCOMES:
Pediatric Quality Of Life score (PedsQL) | Assessed every two weeks from weeks 0 to 8 (or at time of medical clearance if prior to 8 weeks).
  Longitudinal changes in score on the PedsQL questionnaire (Teen;13-19, parent)
Sport Concussion Assessment tool 5 (symptom scores) | Assessed weekly from weeks 0 and 8 (or time of medical clearance to return to sport if prior to 8 weeks)
  Longitudinal changes in symptom scores on the SCAT5 questionnaire ( Teen;13-19, parent)
Adherence to prescribed exercise | Assessed weekly from weeks 0 and 8 (or time of medical clearance if prior to 8 weeks).
  Self reported adherence patterns to youth prescribed home exercise programs
Activity (kcal/day) | 0-8 weeks (or time of medical clearance if prior to 8 weeks)
  Amount of exercise induced (kcal/day) measured using an Actigraph)
Symptom scores on the Sport Concussion Assessment Tool 5 (SCAT5) | 0-8 weeks (or time of medical clearance if prior to 8 weeks)
  The participants will rate their concussion symptoms using the SCAT5 symptom scale before and after every treadmill test to identify clinical symptom characteristics associated with physical exertion (0-132/132 where 0 indicates no symptoms)
Cognitive activity | Up to 8 weeks
  Cognitive activity as measured by the "Cognitive Activity Scale" (0-4/4)
Incidence of Migraines and Headaches | Up to 8 weeks
  Evaluating the incidence of post-injury International Classification of Headache Disorders (ICHD-3) beta defined migraine headaches and psychiatric outcomes in each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schneider, PT, PhD, Principal Investigator — Sport Injury Prevention Research Centre
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Pan Am Sports Medicine Clinic, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No